CLINICAL TRIAL: NCT05812716
Title: A Randomized Controlled Study to Evaluate the Feasibility and Efficacy of an Online Resilience Intervention for Healthcare Professionals ("resiLIR Healthcare Professionals")
Brief Title: "resiLIR Healthcare Professionals": A Psychological Online Intervention to Enhance Resilience in Healthcare Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leibniz-Institut für Resilienzforschung (LIR) gGmbH (Other)
Collaborators: European Regional Development Fund (Other); Ministry of Science and Health of Rhineland-Palatinate, Germany (Unknown); Fraunhofer Institute for Industrial Mathematics ITWM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01_resiLIR_HCP
Record Dates: First submitted 2023-02-27; First posted 2023-04-14 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Resilience

STUDY DESIGN:
Intervention Model Description: Waitlist control design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will gain access to the 6-week online resilience intervention "resiLIR Healthcare Professionals".
  Interventions: Behavioral: resiLIR Healthcare Professionals
- Waitlist control group (No Intervention): Participants will receive the intervention after the first follow up-assessment (3 months post-intervention of the intervention group).

INTERVENTIONS:
Behavioral: resiLIR Healthcare Professionals — Weeks 1 and 2: Theoretical part on stress, resilience, self-care, and self-compassion
  Weeks 3 to 6: Training phase of a weekly introduced practical exercise (reflection on living with ease, self-compassionate body scan, planning of positive activities, self-compassionate letter). This phase additionally includes smartphone reminders to apply the exercises in everyday life.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate an online resilience intervention with healthcare professionals. Participants will receive a 6-week online intervention addressing resilience and stress with a specific focus on self-care and self-compassion. The main question is whether the intervention is effective in increasing resilience.

DETAILED DESCRIPTION:
Background: Healthcare professionals often experience challenging working conditions, e.g., demanding physical work or time-sensitive tasks, which leads to a high risk of stress-associated disorders or burnout. Especially the COVID-19 pandemic as an additional stressor for healthcare highlighted the role of resilience, that is, the ability to maintain or return to good mental health during stress exposure. To promote mental health and resilience in healthcare professionals, previous studies point to self-care and self-compassion as promising factors.

Objectives: The aim of the study therefore is to examine the feasibility and efficacy of a newly developed online intervention with a focus on self-care and self-compassion to foster resilience in healthcare professionals.

Methods: In a waitlist control design, 240 healthcare professionals will take part in the 6-week resilience intervention "resiLIR Healthcare Professionals". The online intervention contains a theoretical part conveying psychoeducational material as well as a training phase including practical exercises and mini-interventions in everyday life. Participants will assess resilience, burnout, and several resilience factors in online surveys pre-, during and post-intervention as well as 3, 6 and 12 months after completion as follow-up assessments.

Implications: The study will contribute to stress and burnout prevention in healthcare professionals through offering a feasible and evidence-based online intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Fluent in German language
* Access to web-enabled devices (tablet/laptop/computer)
* Smartphone with internet access
* Trained and employed as health care professionals

Exclusion Criteria:

* Acute mental health crisis (e.g., suicidality)
* Psychiatric/psychotherapeutic treatment
* Neurodegenerative disease(s)
* Diagnosis of schizophrenia or other psychotic disorders, bipolar disorder, post-traumatic stress disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Change of Resilience measured with stressor reactivity score (Kalisch et al., 2015, 2021) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Stressor reactivity score (Kalisch et al., 2015, 2021): Stressor reactivity can be approximated by relating self-reported mental-health problems to the corresponding stressor exposure within the same timeframe (for scales for mental health problems and stressor exposure, see secondary outcomes). The stressor reactivity (SR) score will be computed as an individual score against normal stressor reactivity (see Kalisch et al., 2021), where normal stressor reactivity is the regression line of average mental health problems against average stressor exposure across all time points in the trial population and one's individual SR score at any time point is the distance to the regression line. The inverse of the SR score is considered an approximative index of outcome-based resilience. Therefore, a lower SR score indicates higher resilience. Change calculated between time points named in time frame, for details, see statistical analysis plan.

SECONDARY OUTCOMES:
Change in Resilience measured with Brief Resilience Scale (BRS; Chmitorz et al., 2018) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Brief Resilience Scale (BRS; Chmitorz et al., 2018):
  Participants rate different items on a scale from 1 to 5. Items 2, 4 and 6 are inverted; scale mean is formed. Higher scores indicate higher resilience. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Mental Health measured with General Health Questionnaire (GHQ-12; Schrnitz et al., 1999) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  General Health Questionnaire (GHQ-12; Schrnitz et al., 1999):
  Participants rate different items on a scale from 0 to 3. Items 14, 15, 10, 16, 18 and 19 are inverted; sum score is formed. Higher scores indicate lower mental health. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Stress measured with Perceived Stress Scale (PSS-2+2; Schäfer et al., in preparation) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Perceived Stress Scale (PSS-2+2; Schäfer et al., in preparation):
  Participants rate different items on a scale from 1 to 5. Items 1 and 2 are inverted; scale mean is formed. Higher scores indicate higher stress. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Well-being measured with WHO-5 Well-Being Index (Brähler et al., 2007) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  WHO-5 Well-Being Index (Brähler et al., 2007):
  Participants rate different items on a scale from 1 to 6. Sum score is formed. Higher scores indicate higher well-being. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Anxiety measured with Generalized Anxiety Disorder-7 (GAD-7; Löwe et al., 2002) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Generalized Anxiety Disorder-7 (GAD-7; Löwe et al., 2002):
  Participants rate different items on a scale from 0 to 3. Sum score is formed. Higher scores indicate higher anxiety. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Depression measured with Patient Health Questionnaire-9 (PHQ-9; Löwe et al., 2002) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Patient Health Questionnaire-9 (PHQ-9; Löwe et al., 2002):
  Participants rate different items on a scale from 0 to 3. Sum score is formed. Higher scores indicate higher depression. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Self Compassion measured with Self-Compassion Scale Deutsch (SCS-D; Hupfeld & Ruffieux, 2011) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Self-Compassion Scale Deutsch (SCS-D; Hupfeld & Ruffieux, 2011):
  Participants rate different items on a scale from 1 to 5. Items 1, 2, 4, 6, 8, 11, 13, 16, 18, 20, 21, 24 and 25 are inverted; scale mean is formed. Higher scores indicate higher self compassion. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Self-care measured with Hamburg Self-Care Survey (Harfst et al., 2009) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Hamburg Self-Care Survey (Harfst et al., 2009):
  Participants rate different items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher self-care. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Mindfulness measured with Mindful Attention and Awareness Scale (MAAS-Short; Höfling et al., 2011) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mindful Attention and Awareness Scale (MAAS-Short; Höfling et al., 2011):
  Participants rate different items on a scale from 1 to 6. Items 1, 2, 3, 4 and 5 are inverted; scale mean is formed. Higher scores indicate higher mindfulness. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Work-Life Balance measured with Trier Short Scale for Assessing Work-life-balance (TKS-WLB; Syrek et al., 2011) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Trier Short Scale for Assessing Work-life-balance (TKS-WLB; Syrek et al., 2011) Participants rate different items on a scale from 1 to 5. Item 2 is inverted. Higher scores indicate higher work-life-balance. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Burnout measured with Maslach Burnout Inventory (MBI-D; Büssing & Perrar, 1992) | baseline (pre), 4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Maslach Burnout Inventory (MBI-D; Büssing & Perrar, 1992):
  Participants rate different items on a scale from 0 to 6. Items 4, 7, 9, 12, 17, 18, 19, 21, 23 and 24 are inverted. Higher scores indicate higher burnout. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change in Optimism measured with Optimism-Pessimism-Scale (SOP-2; Kemper et al., 2014) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Optimism-Pessimism-Scale (SOP-2; Kemper et al., 2014):
  Participants rate different items on a scale from 1 to 7. Item 2 is inverted, scale mean is formed. Higher scores indicate higher optimism. Change calculated between time points named in time frame.
Change in Sense of Coherence measured with Sense of Coherence Scale-29 (SOC-29; Singer et al., 2007) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Sense of Coherence Scale-29 (SOC-29; Singer et al., 2007):
  Participants rate different items on a scale from 1 to 7. Item 2, 5, 6, 7, 8, 12, 14, 15, 17, 21, 24 and 28 are inverted, scale mean is formed. Higher scores indicate higher sense of coherence. Change calculated between time points named in time frame.
Change in Meaning and Purpose measured with Subscale of Comprehensive Inventory of Thriving (CIT; Hausler et al., 2017) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Comprehensive Inventory of Thriving (CIT; Hausler et al., 2017):
  Participants rate different items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher meaning. Change calculated between time points named in time frame.
Change in Acceptance measured with Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011):
  Participants rate different items on a scale from 1 to 6. Scale mean is formed. Higher scores indicate higher acceptance. Change calculated between time points named in time frame.
Change in Positive Reappraisal measured with Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011):
  Participants rate different items on a scale from 1 to 6. Scale mean is formed. Higher scores indicate higher positive reappraisal. Change calculated between time points named in time frame.
Change in Self-Efficacy measured with German Version of Self-Efficacy Short Scale (ASKU; Beierlein et al., 2014) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  German Version of Self-Efficacy Short Scale (ASKU; Beierlein et al., 2014):
  Participants rate different items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher self-efficacy. Change calculated between time points named in time frame.
Change in Social Support measured with Oslo Social Support Scale (OSS-3; Kocalevent et al., 2018) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Oslo Social Support Scale (OSS-3; Kocalevent et al., 2018):
  Participants rate different items on a scale from 1 to 4/ 1 to 5. Sum score is formed. Higher scores indicate higher social support. Change calculated between time points named in time frame.
Change in Positive Appraisal Style (content aspects) measured with Positive Appraisal Style Content (PASS-content) (no publication, pre-version in Petri-Romao et al., 2021) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Positive Appraisal Style Content (PASS-content; no publication, pre-version in Petri-Romao et al., 2021) Participants rate different items on a scale from 1 to 4. Scale mean is formed. Higher scores indicate higher positive appraisal (content aspects). Change calculated between time points named in time frame.
Change in Positive Appraisal Style (procedural aspects) measured with Positive Appraisal Style Content (PASS-process) (no publication, pre-version in Petri-Romao et al., 2021) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Positive Appraisal Style Content (PASS-process) (no publication, pre-version in Petri-Romao et al., 2021) Participants rate different items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher positive appraisal (procedural aspects). Change calculated between time points named in time frame.
Change in Internal and External Locus of Control measured with Internal-External Locus of Control Short Scale-4 (IE-4; Kovaleva et al., 2014) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Internal-External Locus of Control Short Scale-4 (IE-4; Kovaleva et al., 2014):
  Participants rate different items on two subscales from 1 to 5. Scale mean for each subscale is formed. Higher scores on the first subscale indicate higher internal locus of control, higher scores on the second subscale indicate higher external locus of control. Change calculated between time points named in time frame.
Change in Coping measured with Coping Orientation to Problems Experienced Inventory (Brief-COPE; Knoll et al., 2005) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Coping Orientation to Problems Experienced Inventory (Brief-COPE; Knoll et al., 2005):
  Participants rate different items on two subscales from 1 to 4. Scale mean for each subscale is formed. Higher scores on the first subscale indicate higher adaptive coping, higher scores on the second subscale indicate higher maladaptive coping. Change calculated between time points named in time frame.
Change of Self-Esteem measured with German Single-Item Self-Esteem Scale (G-SISE; Brailovskaia & Margraf, 2020) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  German Single-Item Self-Esteem Scale (G-SISE; Brailovskaia & Margraf, 2020):
  Participants rate one item on a scale from 1 to 5. Higher scores indicate higher self-esteem. Change calculated between time points named in time frame.
Positive Affect measured with Subscale of Positive and Negative Affect Schedule (PANAS; Breyer & Bluemke, 2016) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Positive and Negative Affect Schedule (PANAS; Breyer & Bluemke, 2016) Participants rate 10 items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher positive affect. Change calculated between time points named in time frame.
Satisfaction with Life measured with Satisfaction with Life Scale (SWLS; Janke & Glöckner-Rist, 2012) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Satisfaction with Life Scale (SWLS; Janke & Glöckner-Rist, 2012):
  Participants rate 5 items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher satisfaction with life. Change calculated between time points named in time frame.
Functioning measured with World Health Organization Disability Assessment Schedule (WHODAS 2.0; Üstün et al., 2010) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  World Health Organization Disability Assessment Schedule (WHODAS 2.0; Üstün et al., 2010):
  Participants rate 12 items on a scale from 1 to 5. Sum score is formed. Higher scores indicate lower functionality. Change calculated between time points named in time frame.
Coping Flexibility measured with Coping Flexibility Questionnaire Revised (CFQ-R; Kato, 2020) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Coping Flexibility Questionnaire Revised (CFQ-R; Kato, 2020):
  Participants rate 12 items on a scale from 1 to 4. There are three sub scales. Scale mean is formed, respectively. Higher scores indicate higher flexibility. Change calculated between time points named in time frame.
Satisfaction with Intervention (only for the intervention group) measured with Client Satisfaction Questionnaire-Intervention (CSQ-I; Boß et al., 2016) | 6-8 weeks (post)
  Client Satisfaction Questionnaire-Intervention (CSQ-I; Boß et al., 2016):
  Participants rate 8 items on a scale from 1 to 4. Scale mean is formed. Higher scores indicate higher client satisfaction.
Adverse Effects (only for the intervention group) measured with Inventory of Negative Effects of Psychotherapy for Online-Interventions (INEP-ON; Ladwig et al., 2014) | 6-8 weeks (post)
  Inventory of Negative Effects of Psychotherapy for Online-Interventions (INEP-ON; Ladwig et al., 2014): Participants rate in total 23 items. Of these, items 1 to 11 are rated on a 7-point scale ranging from 3 (positive outcome, like "better" or "supportive") to -3 (negative outcome, like "worse" or "disturbing"); items 12 to 21 are rated on a 4-point scale ranging from 0 (fully disagree) to 3 (fully agree) and then rated if a possible change is attributed to the intervention or life circumstances. Items 22 and 23 are also rated on a 4-point scale ranging from 0 (fully disagree) to 3 (fully agree).
  We are not sure whether the questionnaire can be evaluated with a sum score or mean, we have contacted the author about it to receive instructions.
Relationship to Intervention (only for the intervention group) measured with Mobile Agnew Relationship Measure (mARM; von Wulffen et al., 2022) | 6-8 weeks (post)
  Mobile Agnew Relationship Measure (mARM; von Wulffen et al., 2022): Participants rate 24 items on a scale from 1 to 7. Items 4, 8, 16, and 18 are reverse coded. There are 5 sub scales. Scale mean is formed, respectively. Higher scores indicate higher bond/ confidence/ openness/ relationship/ client initiative.
Work Engagement measured with Utrecht Work Engagement Scale (UWES-9; Schaufeli et al., 2006) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Utrecht Work Engagement Scale (UWES-9; Schaufeli et al., 2006): The UWES-9 consists of 9 items which are rated on a 7-point scale ranging from 0 (never) to 6 (always). There are 3 subscales. Scale mean is formed, respectively. Higher scores indicate higher vigor / dedication / absorption. Change calculated between time points named in time frame.
Perceived Occupational Stress measured with Perceived Occupational Stress Scale (Marcatto et al., 2021) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 12 months (second-follow up)
  Perceived Occupational Stress Scale (POS; Marcatto et al., 2021): The POS scale presents four items which are self-reported along a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Their answers are averaged. Higher scores indicate higher perceived occupational stress. Change calculated between time points named in time frame.

OTHER OUTCOMES:
Attitudes towards Psychological Online Interventions measured with Attitudes towards Psychological Online Interventions Questionnaire (APOI; Schröder et al., 2015) | baseline (pre)
  Attitudes towards Psychological Online Interventions Questionnaire (APOI; Schröder et al., 2015):
  Participants rate 16 items on a scale from 1 to 7. There are four sub scales (Scepticism and perception of Risks, Confidence in Effectiveness, Technologization Threat, Anonymity Benefits), scale mean is formed, respectively. Higher scores indicate higher Scepticism, etc..
Personality measured with Big Five Inventory-10 (BFI-10; Rammstedt et al., 2017) | baseline (pre)
  Big Five Inventory-10 (BFI-10; Rammstedt et al., 2017):
  Participants rate 10 items on a scale from 1 to 5. There are five sub scales (Extraversion, Openness, Neuroticism, Agreeableness, Conscientiousness). Scale mean is formed, respectively. Higher scores indicate higher Extraversion, etc.
Sociodemographic Variables | baseline (pre)
  Single Items: age, sex, education
Socioeconomic Variables | baseline (pre)
  number of people living in household, number of children living in household, household net income, individual net income
Change of belief Towards Mental Illness measured with Belief Towards Mental Illness Scale (Hirai & Clum, 2018) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Belief Towards Mental Illness Scale (Hirai & Clum, 2018):
  Participants rate 21 items on a scale from 1 to 6. There are three sub scales (Dangerousness, Poor social and interpersonal skills, Incurability). Scale mean is formed, respectively. Higher scores indicate higher Dangerousness, etc.Change calculated between time points named in time frame.
Change of help-seeking Behavior measured with General Help Seeking Scale (Rickwood et al., 2005) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  General Help Seeking Scale (Rickwood et al., 2005):
  Participants rate 15 items on a scale from 1 to 4. There are three sub scales (level of intention for seeking informal help, level of intention for seeking formal help, level of intention to seek help from no-one). Scale mean is formed, respectively. Higher scores indicate higher level of intention for seeking informal help, etc. Change calculated between time points named in time frame.
Change of help-seeking Behavior measured with Attitudes Toward Seeking Professional Psychological Help (Kessler et al., 2015) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Attitudes Toward Seeking Professional Psychological Help (Kessler et al., 2015): Participants rate 24 items on a scale from 1 to 5. Items 1, 3, 4, 6, 7, 9, 11, 12, 14, 16, 17, 18, 20, 21 and 24 are inverted. There are three sub scales (Psychological Openness, Help-Seeking Propensity, Indifference to stigma). Scale mean is formed, respectively. Higher scores indicate higher level of Psychological Openness, etc. Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with Mental Health Literacy Questionnaire (Dias et al., 2018) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mental Health Literacy Questionnaire (Dias et al., 2018):
  Participants rate 29 items on a scale from 1 to 5. Items 6, 10, 13, 15, 21 and 23 are inverted. Sum score is formed. Higher scores indicate higher health literacy.Change calculated between time points named in time frame.
Change in Mental Health Literacy measured with Mental Health Literacy Scale (O'Connor & Casey, 2015) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mental Health Literacy Scale (O'Connor & Casey, 2015):
  Participants rate 35 items on a scale from 1 to 4/5. Items 10, 12, 15, 20, 21, 22, 23, 24, 25, 26, 27, 28 are inverted. Sum score is formed. Higher scores indicate higher health literacy. Change calculated between time points named in time frame.
Change in Mental Health Literacy measured with Mental Health Knowledge Schedule (Evans-Lacko et al., 2010) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mental Health Knowledge Schedule (Evans-Lacko et al., 2010): Participants rate 6 items on a scale from 1 to 6. Sum score is formed where 6 (don't know) is equalized to a score of 3. Higher scores indicate higher health literacy. Change calculated between time points named in time frame.
Change in Mental Health Literacy measured with Health Literacy Survey EU 16 (Jordan & Hoebel, 2015) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Health Literacy Survey EU 16 (Jordan & Hoebel, 2015) Participants rate 16 items on a scale from 1 to 4. Sum score is formed where 1/2 are summed up to a score of 1 and 3/4 are summed up to a score of 0. Higher scores indicate higher health literacy. Change calculated between time points named in time frame.
Change in Mental Health Literacy measured with eHealth Literacy Scale (Soellner et al., 2014) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  eHealth Literacy Scale (Soellner et al., 2014): Participants rate 8 items on a scale from 1 to 5. There are two subscales (Information seeking/ Information appraisal). Scale mean is formed. Higher scores indicate higher information seeking/ information appraisal. Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with Well-being Literacy Scale (Hou et al., 2021) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Well-being Literacy Scale (Hou et al., 2021): The scale consists of 6 items. Each item is rated on a 7-point Likert scale, from 1 (Strongly disagree) to 7 (Strongly agree). Scale mean is formed. Higher scores indicate higher mental health literacy. Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with STRESS K-10 (Giesinger et al., 2008) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  STRESS K-10 (Giesinger et al., 2008):
  Participants rate 10 items on a scale from 1 to 5. Sum score is formed. Higher scores indicate higher stress. Change calculated between time points named in time frame.
Change of Knowledge of psychosocial care structures measured with Questionnaire to survey knowledge of psychosocial care structures. (Fritz, 2021, in preparation) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Questionnaire to survey knowledge of psychosocial care structures. (Fritz, 2021, in preparation) Participants rate 8 items on a scale from 1 to 3 (yes, no, I don't know). Sum score is formed. Higher scores indicate higher knowledge. Change calculated between time points named in time frame.
Work-related variables | baseline (pre)
  number of working hours according to contract, frequency and amount of working extra hours, leadership responsibility, working (night) shifts.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | baseline (pre)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017):
  Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 4 weeks (intermediate)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017):
  Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 6-8 weeks (post)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017):
  Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 3 months (first follow-up)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017):
  Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 6 months (second follow-up)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017):
  Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 12 months (third follow-up)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017):
  Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Stressors measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | baseline (pre)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020):
  Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Occurrence of Stressors measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 4 weeks (intermediate)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020):
  Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Occurrence of Stressors measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 6-8 weeks (post)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020):
  Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Occurrence of Stressors measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 3 months (first follow-up)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020):
  Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Occurrence of Stressors measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 6 months (second follow-up)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020):
  Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Occurrence of Stressors measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 12 months (third follow-up)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020):
  Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors. Change calculated between time points named in time frame, for details, see statistical analysis plan.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Tüscher, Principal Investigator — Leibniz Institute of Resilience Research
Locations (1):
- Leibniz Institute for Resilience Research gGmbH, Mainz, Rhineland-Palatinate, Germany

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT05812716/SAP_000.pdf